CLINICAL TRIAL: NCT07220759
Title: Efficacy and Safety of Cagrilintide for Weight Management in Participants With Overweight or Obesity and Type 2 Diabetes
Brief Title: Weight Loss in People Living With Overweight or Obesity and Type 2 Diabetes Following Treatment With Cagrilintide
Acronym: RENEW 2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9833-8243; U1111-1314-9328 (Other: World Health Organization (WHO)); 2024-519531-41 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2025-10-23; First posted 2025-10-24 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Overweight; Obesity; Type 2 Diabetes
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2 | interventions — cagrilintide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cagrilintide (Experimental): Participants will receive cagrilintide subcutaneously once weekly for 64 weeks.
  Interventions: Drug: Cagrilintide
- Placebo (Placebo Comparator): Participants will receive placebo matched to cagrilintide subcutaneously once weekly for 64 weeks.
  Interventions: Drug: Placebo (matched to Cagrilintide)

INTERVENTIONS:
Drug: Cagrilintide — Cagrilintide will be administered subcutaneously with a pen-injector as an adjunt to lifestyle intervention counselling.
  Arms: Cagrilintide
Drug: Placebo (matched to Cagrilintide) — Placebo matched to cagrilintide will be administered subcutaneously with a pen-injector as an adjunt to lifestyle intervention counselling.
  Arms: Placebo

SUMMARY:
This study will look at how much cagrilintide helps people with overweight or obesity and type 2 diabetes lower their body weight. Cagrilintide is a new investigational medicine. Doctors may not yet prescribe cagrilintide. Participant will either get cagrilintide or placebo. Which treatment participant get is decided by chance. Participants are two times more likely to get cagrilintide than placebo. Like all medicines, the study medicine may have side effects. For each participant, the study will last for about 1 year and 6 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* Female or male (sex at birth).
* Age 18 years or above at the time of signing the informed consent.
* History of at least one self-reported unsuccessful dietary effort to lose body weight.(a*)
* Body mass index (BMI) >= 27.0 kilogram per square meter (kg/m^2).(a*)
* Diagnosed with type 2 diabetes >= 180 days before screening.
* Treatment with either lifestyle intervention(a*), or:

  * Stable treatment (same drug(s), dose and dosing frequency) for at least 90 days before screening with 1-3 marketed oral antidiabetic drugs (metformin, α-glucosidase inhibitors (AGI), glinides, sodium-glucose cotransporter 2 inhibitor (SGLT2i), thiazolidinediones, Dipeptidyl peptidase-4 inhibitor (DPP-4i) or sulphonylureas (SU) as a single agent or in combination according to local practice.(a*)
  * For up to 30% of participants the following concomitant medication is allowed:

    * Treatment for any indication with a stable dose of glucagon-like peptide-1 (GLP-1) containing medication, stable for at least 1 year before screening (a*) and/or
    * Treatment with basal insulin minimum (0.25 units per kilogram per day (U/kg/day) or 20 units per day [U/day]) stable for at least 90 days before screening.(a*)

Key Exclusion Criteria:

* Treatment, or intention to initiate treatment, with any medication prescribed for the indication of weight management within 180 days before screening.(a*)
* Treatment with glucagon-like peptide-1 (GLP-1) receptor agonist (RA) or GLP-1 containing medication within 180 days before screening, apart from those randomized according to inclusion criteria 7bi.(a*)
* Previous dosing of marketed or non-marketed amylin-based compounds.(a*) (a*) - As declared by the participant, reported in the medical records or at the investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2027-06-09 (Estimated); Study Completion 2027-07-28 (Estimated)

PRIMARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to end of treatment (week 64)
  Measured as percentage (%) of body weight.
Number of participants with achievement of greater than or equals (>=) 5% body weight reduction | From baseline (week 0) to end of treatment (week 64)
  Measured as count of participants.

SECONDARY OUTCOMES:
Number of participants with achievement of >= 10% body weight reduction | From baseline (week 0) to end of treatment (week 64)
  Measured as count of participants.
Number of participants with achievement of >= 15% body weight reduction | From baseline (week 0) to end of treatment (week 64)
  Measured as count of participants.
Change in waist circumference | From baseline (week 0) to end of treatment (week 64)
  Measured as centimeter (cm).
Ratio to baseline in lipids: triglycerides | From baseline (week 0) to end of treatment (week 64)
  Measured as ratio.
Ratio to baseline in high sensitivity C-reactive protein (hsCRP) | From baseline (week 0) to end of treatment (week 64)
  Measured as ratio.
Change in impact of weight on quality of life-lite clinical trials version (IWQOL-Lite-CT) physical function score | From baseline (week 0) to end of treatment (week 64)
  Measured as score on a scale. IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Higher scores indicate better levels of functioning. The physical function score ranges from 0-100.
Change in body weight | From baseline (week 0) to end of treatment (week 64)
  Measured as kilogram (kg).
Change in SF-36v2® health survey acute (SF-36v2® acute) physical component summary score | From baseline (week 0) to end of treatment (week 64)
  Measured as score on a scale. SF-36v2 Acute measures Health-Related Quality of Life (HRQoL). The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2 Acute scores are norm-based scores, that is. transformed to a scale where the 2009 US general population has a mean of 50 and a standard deviation of 10. Higher scores indicate better functional health and well-being. The physical component summary score ranges from 6.1 to 79.7.
Change in SF-36v2® mental component summary score | From baseline (week 0) to end of treatment (week 64)
  Measured as score on a scale. SF-36v2 Acute measures Health-Related Quality of Life (HRQoL). The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2 Acute scores are norm-based scores, that is. transformed to a scale where the 2009 US general population has a mean of 50 and a standard deviation of 10. Higher scores indicate better functional health and well-being. The mental component summary score ranges from -3.8 to 78.7.
Change in IWQOL-Lite-CT total score | From baseline (week 0) to end of treatment (week 64)
  Measured as score on a scale. IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Higher scores indicate better levels of functioning. The total score ranges from 0-100.
Number of participants with achievement of at least 14.6-point increase in IWQOL-Lite-CT physical function score (yes/no) | From baseline (week 0) to end of treatment (week 64)
  Measured as count of participants. IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Higher scores indicate better levels of functioning. The physical function score ranges from 0-100.
Change in systolic blood pressure (SBP) | From baseline (week 0) to end of treatment (week 64)
  Measured as millimeter of mercury (mmHg).
Change in diastolic blood pressure (DBP) | From baseline (week 0) to end of treatment (week 64)
  Measured as mmHg.
Ratio to baseline in lipids: total cholesterol | From baseline (week 0) to end of treatment (week 64)
  Measured as ratio.
Ratio to baseline in lipids: high-density lipoprotein (HDL) cholesterol | From baseline (week 0) to end of treatment (week 64)
  Measured as ratio.
Ratio to baseline in lipids: low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to end of treatment (week 64)
  Measured as ratio.
Ratio to baseline in lipids: very low-density lipoprotein (VLDL) cholesterol | From baseline (week 0) to end of treatment (week 64)
  Measured as ratio.
Ratio to baseline in lipids: non-HDL cholesterol | From baseline (week 0) to end of treatment (week 64)
  Measured as ratio.
Ratio to baseline in lipids: free fatty acids | From baseline (week 0) to end of treatment (week 64)
  Measured as ratio.
Change in glycated haemoglobin (HbA1c) in percentage-points (%-points) | From baseline (week 0) to end of treatment (week 64)
  Measured as %-points.
Change in HbA1c in millimole per mole (mmol/mol) | From baseline (week 0) to end of treatment (week 64)
  Measured as mmol/mol.
Change in fasting plasma glucose (FPG) in millimole per liter (mmol/L) | From baseline (week 0) to end of treatment (week 64)
  Measured as mmol/L.
Change in FPG in milligram per deciliter (mg/dL) | From baseline (week 0) to end of treatment (week 64)
  Measured as mg/dL.
Ratio to baseline in fasting serum insulin | From baseline (week 0) to end of treatment (week 64)
  Measured as ratio.
Number of treatment emergent adverse events | From baseline (week 0) to end of study (week 71)
  Measured as count of events.
Number of treatment emergent serious adverse events (TESAEs) | From baseline (week 0) to end of study (week 71)
  Measured as count of events.
Number of clinically significant hypoglycaemic episodes (level 2):<3.0 mmol/L [54 mg/dL], confirmed by blood glucose meter | From baseline (week 0) to end of study (week 71)
  Measured as count of events.
Number of severe hypoglycaemic episodes (level 3): hypoglycaemia associated with severe cognitive impairment requiring external assistance for recovery, with no specific glucose threshold | From baseline (week 0) to end of study (week 71)
  Measured as count of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency' (dept. 2834), Study Director — Novo Nordisk A/S
Locations (67):
- United States (21):
  - Univ of Alabama_Birmingham, Birmingham, Alabama
  - Chambliss Clinical Trials, LLC, Montgomery, Alabama
  - Elite Clinical Network - Tucson, Tucson, Arizona
  - Scripps Whittier Diabetes Inst, La Jolla, California
  - Clinical Trials Research, Lincoln, California
  - Pacific Clinical Studies, Los Alamitos, California
  - Walgreens - Store 4442, Kissimmee, Florida
  - Optimal Research Sites, Orange City, Florida
  - Center for Diab,Obes & Metab, Pembroke Pines, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - East West Med Res Inst, Honolulu, Hawaii
  - MediSphere Medical RC, Evansville, Indiana
  - Walgreens - Store 3915, Las Vegas, Nevada
  - Chear Center LLC, The Bronx, New York
  - Centricity Res New Bern, New Bern, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Holston Medical Group_Bristol, Bristol, Tennessee
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - TPMG Clinical Research, Newport News, Virginia
  - National Clin Res Inc., Richmond, Virginia
- Argentina (3):
  - Buenos Aires Mácula, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - CICEMO- Consultorio de Investigación Clínica EMO, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Centro Medico Dra. Laura Maffei e Investigacion Clínica Apli, Buenos Aires
- Canada (9):
  - OCT Research ULC (dba Okanagan Clinical Trials), Kelowna, British Columbia
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Nova Scotia Hlth Halifax, Halifax, Nova Scotia
  - Centricity Research Brampton Endocrinology, Brampton, Ontario
  - Hamilton Medical Rsrch Grp, Hamilton, Ontario
  - Wharton Med Clin Trials, Hamilton, Ontario
  - Milestone Research, London, Ontario
  - Centricity Res Pointe-Claire, Pointe-Claire, Quebec
  - Diex Recherche Victoriaville, Victoriaville, Quebec
- Croatia (4):
  - Opca bolnica Karlovac, Karlovac
  - Specijalna Bolnica za medicinsku rehabilitaciju Krapinske Toplice_Endocrinology, Krapinske Toplice
  - Poliklinika SLAVONIJA OSIJEK, Osijek
  - Poliklinika Solmed, Zagreb
- Czechia (3):
  - Lékařský dům Géčko, České Budějovice
  - Milan Kvapil s.r.o., Prague
  - EUC Klinika Praha a.s., Prague
- Hungary (4):
  - Debreceni Egyetem, Debrecen, Hajdú-Bihar
  - QUALICLINIC Egészségügyi Szolgáltató és Kutatásszervező Kft, Budapest, Pest County
  - Óbudai Egészségügyi Centrum, Budapest, Pest County
  - Komáromi Selye János Kórház, Komárom
- Romania (5):
  - Diabmed Dr Popescu Alexandrina SRL, Ploieşti, Prahova
  - CMI Dr. Pletea Noemi SRL, Bacau
  - Diabet Med SRL, Bucharest
  - S.C Milena Sante SRL, Galati
  - Clinica Korall S.R.L. Satu Mare, Satu Mare
- Slovakia (3):
  - Nemocnica akademika L. Derera, UNB, Bratislava
  - DIAB s.r.o., Rožňava
  - IRIDIA s.r.o., Vrútky
- South Korea (6):
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - The Catholic University of Korea, Yeouido ST. Mary's Hospital, Seoul
  - Kyunghee University Medical Center, Seoul
- Switzerland (4):
  - Universitätsspital Basel, Basel
  - Centre hospitalier universitaire vaudois CHUV, Lausanne
  - Kantonsspital Olten, Olten
  - Diabetes Adipositas Zentrum Zürich, Zollikerberg
- United Kingdom (5):
  - Oak Tree Surgery, Liskeard, Cornwall
  - North Coast Medical Ltd, Newquay, Cornwall
  - Brunel Medical Practice, Torquay, Devon
  - Attenborough Surgery, Bushey, Hertfordshire
  - Hammersmith and Fulham Partnership Research Unit - Richford Gate Primary Care Centre, London

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com